CLINICAL TRIAL: NCT02035267
Title: A Multicenter, Double-blind, Placebo-controlled Safety Study of ATX-101 (Deoxycholic Acid) Injection for the Reduction of Localized Subcutaneous Fat in the Submental Area in Subjects With Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) Grade 1 or CR-SMFRS Grade 4
Brief Title: Safety Study of ATX-101 (Deoxycholic Acid) in Subjects With Mild or Extreme Fullness of Submental Fat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATX-101-13-27
Record Dates: First submitted 2014-01-12; First posted 2014-01-14 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-01

CONDITIONS: Moderate to Severe Convexity of Submental Fat; Safety; Efficacy
MeSH Terms: interventions — Deoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo - Grade 1 (Placebo Comparator): Participants received placebo administered in 0.2 mL subcutaneous (SC) injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments. Participants With CR SMFRS Grade 1 (mild).
  Interventions: Drug: Placebo
- ATX-101 deoxycholic acid injection - Grade 1 (Experimental): Participants received deoxycholic acid 2 mg/cm^2 administered in 0.2 mL SC injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments. Participants With Clinician-Reported Submental Fat Rating Scale (CR SMFRS) Grade 1 (mild).
  Interventions: Drug: Deoxycholic Acid
- Placebo - Grade 4 (Placebo Comparator): Participants received placebo administered in 0.2 mL SC injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments. Participants With CR SMFRS Grade 4 (extreme).
  Interventions: Drug: Placebo
- ATX-101 deoxycholic acid injection - Grade 4 (Experimental): Participants received deoxycholic acid 2 mg/cm^2 administered in 0.2 mL SC injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments. Participants with CR SMFRS Grade 4 (extreme).
  Interventions: Drug: Deoxycholic Acid

INTERVENTIONS:
Drug: Deoxycholic Acid — Formulated as an injectable solution containing deoxycholic acid at a concentration of 10 mg/mL.
  Other Names: ATX-101 deoxycholic acid injection
  Arms: ATX-101 deoxycholic acid injection - Grade 1; ATX-101 deoxycholic acid injection - Grade 4
Drug: Placebo — Phosphate buffered saline placebo for injection.
  Arms: Placebo - Grade 1; Placebo - Grade 4

SUMMARY:
The objectives of this study are to explore the safety and efficacy of subcutaneous injections of Deoxycholic Acid relative to placebo, in the submental area in patients with mild or extreme fullness of the submental fat and ratings of 1 or 4.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 18 to 65 years old
* Stable Body weight
* Body Mass Index (BMI) of ≤40.0 kg/m^2
* Acceptable volume of submental fat graded by clinician
* Dissatisfaction with the submental area expressed by the subject
* Signed informed consent form (ICF)
* SMF ratings of 1 or 4

Exclusion Criteria:

* No prior intervention for submental fat (SMF) (eg, liposuction, surgery, or lipolytic agents)
* Presence of clinically significant health problems
* History of trauma associated with the chin or neck areas that in the judgment of the investigator may affect evaluation of safety or efficacy of treatment
* Body mass index ≤40 kg/m^2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Beddingfield, III, MD, PhD, Study Director — Sponsor GmbH
Locations (8):
- United States (8):
  - Newport Beach, California
  - San Francisco, California
  - West Hollywood, California
  - Boca Raton, Florida
  - Coral Gables, Florida
  - Glenn Dale, Maryland
  - Chestnut Hill, Massachusetts
  - St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 61 subjects in the ATX-101 group and 32 subjects in the placebo group, who were further stratified by baseline Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) (grade 1 included 31 ATX-101 and 16 placebo subjects; grade 4 included 30 ATX-101 and 16 placebo subjects).
Groups:
- ATX-101 (Deoxycholic Acid) Injection - Grade 1: Participants with Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) score of 1 (mild submental convexity) received deoxycholic acid 2 mg/cm^2 administered in 0.2 mL subcutaneous (SC) injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
- Placebo Injection - Grade 1: Participants with Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) score of 1 (mild submental convexity) received placebo administered in 0.2 mL subcutaneous (SC) injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
- ATX-101 (Deoxycholic Acid) Injection - Grade 4: Participants with Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) score of 4 (extreme submental convexity) received deoxycholic acid 2 mg/cm^2 administered in 0.2 mL subcutaneous (SC) injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
- Placebo Injection - Grade 4: Participants with Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) score of 4 (extreme submental convexity) received placebo administered in 0.2 mL subcutaneous (SC) injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
Period: Overall Study
Arm/Group | ATX-101 (Deoxycholic Acid) Injection - Grade 1 | Placebo Injection - Grade 1 | ATX-101 (Deoxycholic Acid) Injection - Grade 4 | Placebo Injection - Grade 4
Started | 31 | 16 | 30 | 16
Completed | 31 | 15 | 28 | 15
Not Completed | 0 | 1 | 2 | 1
Not completed — Withdrawal consent-subject convenience | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Other unspecified | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ATX-101 (Deoxycholic Acid) Injection - Grade 1 | Placebo Injection - Grade 1 | ATX-101 (Deoxycholic Acid) Injection - Grade 4 | Placebo Injection - Grade 4 | Total
Number analyzed (Participants) | 31 | 16 | 30 | 16 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (9.68) | 48.4 (8.75) | 52.1 (7.94) | 50.1 (11.21) | 50.0 (9.27)
Age, Customized [Count of Participants; unit: Participants]
  18-30 years | 3 | 1 | 0 | 1 | 5
  31-40 years | 1 | 2 | 4 | 2 | 9
  41-50 years | 16 | 6 | 10 | 5 | 37
  51-65+ years | 11 | 7 | 16 | 8 | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 16 | 25 | 8 | 78
  Male | 2 | 0 | 5 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10 | 6 | 26
  Not Hispanic or Latino | 24 | 13 | 20 | 10 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 3 | 3 | 3 | 1 | 10
  White | 26 | 12 | 27 | 14 | 79
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Fitzpatrick skin type [Count of Participants; unit: Participants] — Fitzpatrick skin type is a numerical classification schema for different skin types and tanning abilities. TYPE 1: Pale white skin, blue/hazel eyes, blond/red hair, always burns, never tans. TYPE 2: Fair skin, blue eyes, burns easily, tans poorly. TYPE 3: Darker white skin, tans after initial burn. TYPE 4: Light brown skin, burns minimally, tans easily. TYPE 5: Brown skin, rarely burns, tans darkly easily. TYPE 6: Dark brown or black skin, never burns, always tans darkly.
  Participants
    I | 2 | 0 | 0 | 0 | 2
    II | 1 | 2 | 9 | 5 | 17
    III | 12 | 6 | 6 | 4 | 28
    IV | 13 | 5 | 9 | 3 | 30
    V | 3 | 2 | 3 | 4 | 12
    VI | 0 | 1 | 3 | 0 | 4
Weight [Mean (Standard Deviation); unit: kg] | 68.22 (12.935) | 67.76 (9.858) | 87.51 (12.009) | 92.23 (17.518) | 78.49 (16.759)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.60 (4.529) | 24.96 (2.928) | 32.46 (3.898) | 31.83 (4.649) | 28.44 (5.547)
BMI category [Count of Participants; unit: Participants]
  30 kg/m^2 or less | 29 | 15 | 9 | 6 | 59
  Greater than 30 kg/m^2 | 2 | 1 | 21 | 10 | 34
Patient-Reported Submental Fat Rating Scale (PR-SMFRS) score [Count of Participants; unit: Participants] — The participant evaluated their chin and neck area using the Patient-Reported Submental Fat Rating Scale (a 5-point scale) where: 0=no chin fat at all (best) to 4= a very large amount of chin fat (worst).
  Participants
    1 | 15 | 6 | 0 | 0 | 21
    2 | 13 | 10 | 5 | 2 | 30
    3 | 2 | 0 | 17 | 8 | 27
    4 | 1 | 0 | 8 | 6 | 15
Submental Skin Laxity Grade (SMSLG) [Count of Participants; unit: Participants] — The SMSLG is an integration of three features: skin wrinkling, adherence to underlying neck structures (bone and muscle) and redundancy (horizontal and vertical folds). Each grade (1=none, 2=mild, 3=moderate and 4=severe) defines the maximal allowed limit for skin wrinkling, adherence to underlying structures and redundancy.
  Participants
    None/mild | 26 | 14 | 20 | 12 | 72
    Moderate/severe | 5 | 2 | 10 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least a 1-Grade Reduction (Improvement) at 12 Weeks From Last Treatment Based on Both the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) and Patient-Reported Submental Fat Rating Scale (PR-SMFRS) Assessments
Description: The investigator evaluated the participant's chin and neck area using the Clinician-Reported Submental Fat Rating Scale (a 5-point scale) where: 0=absent submental convexity (best) to 4= extreme submental convexity (worst).
  The participant evaluated their chin and neck area using the Patient-Reported Submental Fat Rating Scale (a 5-point scale) where: 0=no chin fat at all (best) to 4= a very large amount of chin fat (worst).
Time Frame: Baseline and up to Week 32 (12 weeks after last treatment)
Population: Intent to treat (ITT) population included all randomized participants, whether or not they received the assigned study drug.
Measure: Number; unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection - Grade 1 | Placebo Injection - Grade 1 | ATX-101 (Deoxycholic Acid) Injection - Grade 4 | Placebo Injection - Grade 4
Number analyzed (Participants) | 31 | 15 | 28 | 15
percentage of participants | 61.3 | 6.7 | 89.3 | 13.3

2. Primary Outcome: Percentage of Participants With at Least a 2-Grade Reduction (Improvement) at 12 Weeks From Last Treatment Based on Both the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) and Patient-Reported Submental Fat Rating Scale (PR-SMFRS) Assessments
Description: as for outcome 1
Time Frame: Baseline and up to Week 32 (12 weeks after last treatment)
Population: Intent to treat (ITT) population included all randomized participants, whether or not they received the assigned study drug. Only subjects with baseline CR-SMFRS grade 4 were included, since a 2-grade improvement was not possible for subjects with baseline CR-SMFRS grade 1.
Measure: Number; unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection - Grade 4 | Placebo Injection - Grade 4
Number analyzed (Participants) | 28 | 15
percentage of participants | 42.9 | 0

3. Primary Outcome: Percentage of Participants With at Least a 1-Grade Reduction (Improvement) at 12 Weeks From Last Treatment Based on the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS)
Description: The investigator evaluated the participant's chin and neck area using the CR-SMFRS 5-point scale where: 0=absent submental convexity (best) to 4= extreme submental convexity (worst).
Time Frame: Baseline and up to Week 32 (12 weeks after last treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection - Grade 1 | Placebo Injection - Grade 1 | ATX-101 (Deoxycholic Acid) Injection - Grade 4 | Placebo Injection - Grade 4
Number analyzed (Participants) | 31 | 15 | 28 | 15
percentage of participants | 74.2 | 20.0 | 96.4 | 26.7

4. Primary Outcome: Percentage of Participants With at Least a 2-Grade Reduction (Improvement) at 12 Weeks From Last Treatment Based on the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS)
Description: as for outcome 3
Time Frame: Baseline and up to Week 32 (12 weeks after last treatment)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection - Grade 4 | Placebo Injection - Grade 4
Number analyzed (Participants) | 28 | 15
percentage of participants | 71.4 | 13.3

5. Primary Outcome: Percentage of Participants With at Least a 1-Grade Reduction (Improvement) at 12 Weeks From Last Treatment Based on Patient-Reported Submental Fat Rating Scale (PR-SMFRS)
Description: The participant evaluated their chin and neck area using the PR-SMFRS 5-point scale where: 0=no chin fat at all (best) to 4= a very large amount of chin fat (worst).
Time Frame: Baseline and up to Week 32 (12 weeks after last treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection - Grade 1 | Placebo Injection - Grade 1 | ATX-101 (Deoxycholic Acid) Injection - Grade 4 | Placebo Injection - Grade 4
Number analyzed (Participants) | 31 | 15 | 28 | 15
percentage of participants | 67.7 | 33.3 | 89.3 | 46.7

6. Primary Outcome: Percentage of Participants With at Least a 2-Grade Reduction (Improvement) at 12 Weeks From Last Treatment Based on Patient-Reported Submental Fat Rating Scale (PR-SMFRS)
Description: as for outcome 5
Time Frame: Baseline and up to Week 32 (12 weeks after last treatment)
Population: Intent to treat (ITT) population included all randomized participants, whether or not they received the assigned study drug. Only subjects with baseline CR-SMFRS grade = 4 were included, since a 2-grade improvement was not anticipated for baseline CR-SMFRS grade = 1 subjects.
Measure: Number; unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection - Grade 4 | Placebo Injection - Grade 4
Number analyzed (Participants) | 28 | 15
percentage of participants | 60.7 | 20.0

7. Primary Outcome: Change From Baseline in Submental Skin Laxity Grade Scale (SMSLG)
Description: The SMSLG is an integration of three features: skin wrinkling, adherence to underlying neck structures (bone and muscle) and redundancy (horizontal and vertical folds). Each grade (1=none, 2=mild, 3=moderate and 4=severe) defines the maximal allowed limit for skin wrinkling, adherence to underlying structures and redundancy.
Time Frame: Baseline and up to Week 32 (12 weeks after last treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ATX-101 (Deoxycholic Acid) Injection - Grade 1 | Placebo Injection - Grade 1 | ATX-101 (Deoxycholic Acid) Injection - Grade 4 | Placebo Injection - Grade 4
Number analyzed (Participants) | 31 | 15 | 28 | 15
scores on a scale | -0.3 (0.60) | -0.1 (0.35) | -0.3 (0.55) | -0.2 (0.56)

ADVERSE EVENTS:
Time Frame: Up to 32 Weeks
Description: Safety population included all randomized participants who received at least 1 injection of study drug.
Arm/Group | ATX-101 (Deoxycholic Acid) Injection - Grade 1 | Placebo Injection - Grade 1 | ATX-101 (Deoxycholic Acid) Injection - Grade 4 | Placebo Injection - Grade 4
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/16 | 0/30 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/16 | 1/30 | 0/16
Other Adverse Events (participants affected / at risk) | 30/31 | 15/16 | 29/30 | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | ATX-101 (Deoxycholic Acid) Injection - Grade 1 (N=31) | Placebo Injection - Grade 1 (N=16) | ATX-101 (Deoxycholic Acid) Injection - Grade 4 (N=30) | Placebo Injection - Grade 4 (N=16)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/29 (0) | 0 (0) | 1/25 (1) | 0/8 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | ATX-101 (Deoxycholic Acid) Injection - Grade 1 (N=31) | Placebo Injection - Grade 1 (N=16) | ATX-101 (Deoxycholic Acid) Injection - Grade 4 (N=30) | Placebo Injection - Grade 4 (N=16)
Injection site pain (General disorders) | 23 (82) | 8 (16) | 16 (78) | 5 (19)
Injection site bruising (General disorders) | 15 (35) | 8 (14) | 18 (35) | 9 (16)
Injection site anaesthesia (General disorders) | 15 (16) | 1 (1) | 16 (22) | 1 (2)
Injection site oedema (General disorders) | 13 (34) | 4 (17) | 14 (37) | 3 (11)
Injection site swelling (General disorders) | 13 (20) | 2 (7) | 14 (25) | 2 (2)
Injection site nodule (General disorders) | 4 (4) | 0 (0) | 4 (6) | 0 (0)
Injection site pruritus (General disorders) | 4 (4) | 1 (1) | 3 (4) | 2 (2)
Injection site induration (General disorders) | 4 (4) | 0 (0) | 3 (3) | 1 (1)
Injection site erythema (General disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (3) | 3 (6) | 1 (1)
Skin tightness (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0) | 4 (4) | 0 (0)
Injection site paraesthesia (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site warmth (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/29 (0) | 0 (0) | 0/25 (0) | 1/8 (1)
Cutis laxa (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.